CLINICAL TRIAL: NCT00623558
Title: A Randomized, Multicenter, Open Phase II Study of Cetuximab With Docetaxel, Cisplatin as Induction Chemotherapy in Unresectable, Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Cetuximab as Induction Treatment in Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Clinical Research Center for Solid Tumor, Korea (Other)
Responsible Party: Principal Investigator, Dae Seog Heo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRCST-L0002
Record Dates: First submitted 2008-02-17; First posted 2008-02-26 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-04

CONDITIONS: Head and Neck Neoplasm
Keywords: head and neck neoplasm; cetuximab; docetaxel; cisplatin; radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Docetaxel+CDDP
  Interventions: Drug: Docetaxel; Drug: Cisplatin
- 2 (Experimental): Docetaxel+CDDP+Cetuximab
  Interventions: Drug: Cetuximab; Drug: Docetaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Cetuximab — 400 mg/m2 first dose, then 250 mg/m2 weekly for 9 weeks
  Arms: 2
Drug: Docetaxel — 75 mg/m2, day 1 of every 3 weeks for 9 weeks (3 cycles)
Drug: Cisplatin — 75 mg/m2, day 1 of every 3 weeks for 9 weeks (3 cycles)

SUMMARY:
The aim of the study is to investigate the efficacy and safety of cetuximab, docetaxel, cisplatin combination as induction therapy in locally advanced head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, locally advanced (cT4b &/or cN2-3) HNSCC
* ECOG performance status 0-1
* Age 18 or older than 18 years
* Measurable disease by RECIST criteria
* Having signed informed consent
* ALT and AST<2.5 times ULN
* Serum albumin level ≥3.0g/dL
* Serum AKP < 2.5 times ULN
* Bilirubin level < 1.5mg/dL
* Serum creatinine <1.5 times ULN
* WBC>3000/mm3, absolute neutrophil count ≥1500/mm3, platelet>75,000/mm3, Hb>9g/dl

Exclusion Criteria:

* Previous cytotoxic chemotherapy for HNSCC
* Radiotherapy for targeted lesions within six months
* Previous EGFR pathway-targeting therapy
* Prior surgery for cancer (excluding diagnostic biopsy within 4 weeks prior to study entry)
* Distant metastatic disease
* Heart failure, coronary artery disease, myocardial infarction within the last 6 months
* Known allergy to any study treatment
* Pregnancy or lactation period
* Any investigational agent within the past 28 days
* Other previous malignancy within 5 year, except adequately treated in situ cervical cancer, or non-melanoma skin cancer
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-04; Primary Completion 2012-11 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Response rate | after induction treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dae Seog Heo, Prof., Principal Investigator — Clinical Research Center for Solid Tumors, Korea
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee KW, Koh Y, Kim SB, Shin SW, Kang JH, Wu HG, Sung MW, Keam B, Kim DW, Kim TM, Kim KH, Kwon TK, Hah JH, Kim IA, Ahn SH, Yoon DH, Lee SW, Kim SY, Nam SY, Jung KY, Baek SK, Hong SH, Lee SH, Heo DS. A Randomized, Multicenter, Phase II Study of Cetuximab With Docetaxel and Cisplatin as Induction Chemotherapy in Unresectable, Locally Advanced Head and Neck Cancer. Oncologist. 2015 Oct;20(10):1119-20. doi: 10.1634/theoncologist.2015-0208. Epub 2015 Aug 24. PMID 26304911